CLINICAL TRIAL: NCT03470597
Title: Registry Study on Effect of Excessive Iodine Exposure on Maternal and Fetal Outcomes
Brief Title: Registry Study for Pregnant Women With Iodine Overload
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Rongrong Li, nutrition physician, Peking Union Medical College Hospital
Other Study IDs: Liuyanping2
Record Dates: First submitted 2018-02-06; First posted 2018-03-20 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Iodine Overload in Pregnancy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women with pre-gestational HSG history: All enrolled pregnant women with pre-gestational ethiodized-oil HSG will be followed up without grouping and be kept track for maternal and offspring's health outcomes in this case registry study.
  Interventions: Other: dietary iodine restriction on subjects with iodine overload

INTERVENTIONS:
Other: dietary iodine restriction on subjects with iodine overload — In this case registry study (observational study),all intervention will be performed not for research purposes, but only part of routine treatment, which will be recorded in database of the registry study.

SUMMARY:
Pre-gestational performance of hysterosalpingography (HSG) using an oil-soluble iodinated contrast medium has been demonstrated to be the main cause of excessive iodine exposure for pregnant women. However, its long-term health effects on the mothers and offsprings have not been adequately elucidated. A case registry study is designed to follow up all the pregnant women with pre-gestational history of ethiodized-oil HSG examination and try to keep track of maternal and fetal outcomes.

ELIGIBILITY:
Inclusion Criteria:

Must be pregnant when enrolled in this study. Must have undergone examination of ethiodized-oil HSG before this pregnancy. Clinical diagnosis of iodine excess (with the mean urine iodine concentration ≥250μg/L and the serum iodine concentration >92μg/L).

Exclusion Criteria:

Having past history of partial or total resection of thyroid glands. Having medical history of thyroid dysfunction before ethiodized-oil HSG examination.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women with excessive iodine exposure caused by pre-gestational ethiodized-oil HSG
Sampling Method: Non-Probability Sample
Enrollment: 195 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
comprehensive pregnant outcomes_prevalence of gestational diabetes | during the whole pregnancy, from date of verification of pregnancy until the date of termination of pregnancy, assessed up to 10 months
  prevalence of gestational diabetes
comprehensive pregnant outcomes_prevalence of gestational hypertension | during the whole pregnancy, from date of verification of pregnancy until the date of termination of pregnancy, assessed up to 10 months
  prevalence of gestational hypertension
comprehensive pregnant outcomes_prevalence of abnormal pregnancy | during the whole pregnancy, from date of verification of pregnancy until the date of termination of pregnancy, assessed up to 10 months
  prevalence of abnormal pregnancy (stillbirth, abortion, premature delivery)
comprehensive pregnant outcomes_rate of cesarean section | at the time of delivery
  rate of cesarean section
comprehensive neonatal outcomes at delivery | at the time of delivery
  Apgar scores of neonates
comprehensive neonatal outcomes_neonatal weight | at the time of delivery
  birth weight of neonates
comprehensive neonatal outcomes_neonatal head circumference | at the time of delivery
  head circumference of neonates
comprehensive neonatal outcomes_neonatal height | at the time of delivery
  height of neonates
comprehensive neonatal outcomes_neonatal BMI | at the time of delivery
  BMI of neonates
comprehensive neonatal outcomes_prevalence of macrosomia or underweight | at the time of delivery
  prevalence of macrosomia or underweight
offspring outcomes_prevalence of thyroid dysfunction | from birth to age of 1 year old, assessed every 6 months
  prevalence of thyroid dysfunction (hyperthyroidism or hypothyroidism)
offspring outcomes_neurodevelopment evaluation in long term | from birth to age of 1 year old, assessed every 6 months
  Norwegian version of the Ages and Stages Questionnaire (ASQ) scores for evaluation of infant neurodevelopment
comprehensive offspring outcomes in long term - weight evaluation | from birth to age of 1 year old, assessed every 3-6 months
  weight of offsprings
comprehensive offspring outcomes in long term - height evaluation | from birth to age of 1 year old, assessed every 3-6 months
  height of offsprings
comprehensive offspring outcomes in long term - BMI evaluation | from birth to age of 1 year old, assessed every 3-6 months
  BMI of offsprings

SECONDARY OUTCOMES:
prevalence of thyroid dysfunction in pregnancy | during the whole pregnancy, from date of verification of pregnancy until the date of termination of pregnancy, assessed up to 10 months
  evaluation of maternal TSH, T3, T4, FT3, FT4, TRAb,Tg-Ab, TPO-Ab
prevalence of iodine overload in neonates | within 1 week after birth of neonates
  prevalence of infants with urinary iodine concentration ≥200μg/L

IPD SHARING:
Plan to Share IPD: No